CLINICAL TRIAL: NCT07140198
Title: Prospective Study to Evaluate the Effectiveness of Hyperbaric Oxygen Therapy (HBOT) to Increase the Survival of Autologous Fat Transfer for Breast Reconstruction After Radiotherapy: A Randomized Controlled Phase II Cross-over Trial
Brief Title: Hyperbaric Oxygen Therapy to Improve Autologous Fat Graft Intake in Irradiated Breast
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Dominik André-Lévigne, Doctor, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-D0050
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Breast Reconstruction; Lipofilling; Hyperbaric Oxygen Therapy
Keywords: breast reconstruction; Irradiation; hyperbaric oxygen therapy; lipofilling
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Other): AFT alone (control) followed by AFT + HBOT (intervention)
  Interventions: Procedure: Hyperbaric Oxygen Therapy; Other: Control
- Sequence BA (Other): AFT + HBOT followed by AFT alone
  Interventions: Procedure: Hyperbaric Oxygen Therapy; Other: Control

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — HBOT will be administered in five sessions (1 on Day 0, 2 on Day 1, 2 on Day 2), beginning immediately after the lipofilling. Each session consists of 100% oxygen inhalation at 2.5 ATA for 90 minutes. Postoperative MRI will be performed six months after each AFT session to assess the volume of retained graft.
Other: Control — Patients in the control group will undergo standard follow-up after the lipofilling without HBOT.

SUMMARY:
The goal of this clinical trial is to learn if hyperbaric oxygen therapy (HBOT) enhances fat graft survival in lipofilling procedures in irradiated breast cancer patients. The main questions it aims to answer are:

Does it improve fat graft survival ? Evaluate safety and tolerability of HBOT in this setting? Researchers will compare patient receiving HBOT to a control group without HBOT to see if.

Sixteen female patients will undergo two autologous fat grafting sessions: one with HBOT and one without, in a randomized sequence. Patients will undergo three MRI during the study to evaluate the fat retention rate.

DETAILED DESCRIPTION:
This is a prospective, monocentric, randomized controlled phase II crossover clinical trial designed to evaluate the efficacy and safety of hyperbaric oxygen therapy (HBOT) in improving fat graft retention following autologous fat transfer (AFT) in breast reconstruction for patients with prior radiotherapy.

AFT is widely used in breast reconstruction but is often less effective in irradiated tissues due to reduced vascularization and oxygenation, which compromises graft survival. HBOT, which involves breathing 100% oxygen at 2.5 atmospheres absolute (ATA), has been shown to promote angiogenesis and tissue oxygenation, potentially improving fat graft integration and reducing complications in irradiated tissues.

The study will enroll 16 adult female patients who have undergone radiotherapy as part of their breast cancer treatment and are scheduled to receive two sessions of AFT. Each participant will be randomized to one of two sequences:

* Sequence AB: AFT alone (control) followed by AFT + HBOT (intervention)
* Sequence BA: AFT + HBOT followed by AFT alone HBOT will be administered in five sessions (1 on Day 0, 2 on Day 1, 2 on Day 2), beginning immediately after the fat grafting procedure. Each session consists of 100% oxygen inhalation at 2.5 ATA for 90 minutes. Postoperative MRI will be performed six months after each AFT session to assess the volume of retained graft.

Primary Objective:

To determine whether HBOT significantly improves fat graft retention in irradiated breast tissue, assessed as the percentage of volume retained (measured by MRI) six months postoperatively.

Secondary Objectives:

* To assess the absolute fat volume retention in milliliters
* To evaluate the safety and tolerability of HBOT in this setting
* To assess the incidence of clinical and radiological complications (e.g., infection, hematoma, oil cysts, liponecrosis) The crossover design minimizes inter-patient variability by allowing each patient to serve as her own control. Randomization occurs immediately after the first AFT session.

The anticipated duration of participation per subject is approximately 12 to 18 months, and the total study duration is estimated at 3 years (from November 2025 to November 2028).

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 y.o. or more) female patients considered for lipofilling following breast reconstruction in an oncological setting which received radiation therapy on the affected breast.
* Ability to provide informed consent, documented by signature

Exclusion Criteria:

* Pregnancy or breastfeeding
* Unability to provide informed consent
* Previous enrolment into the current investigation

Contra-indication to HBOT :

* Anamnestically reported spontaneous pneumothorax
* Status post-thoracotomy
* Significant intra-pulmonary lesions (including emphysematous bullae)
* Respiratory function disorders (both obstructive and restrictive syndromes)
* Pregnancy
* Major psychiatric disorders
* Uncontrollable claustrophobic reaction
* Seizures, even if treated and asymptomatic for some time
* Status post-severe traumatic brain injury with neurological deficits and seizures
* Decompensated heart failure
* Recent myocardial infarction (<6 months) or with persistent hemodynamic sequelae
* Spastic coronary angina
* Cardiac arrhythmias, atrioventricular block, Wolff-Parkinson-White syndrome, sinus node dysfunction, Lown-Ganong-Levine syndrome
* Cardiac pacemakers with unknown pressure resistance
* Severe bradycardia
* Sinus ostium displacement (acute or chronic)
* Displacement of the auditory canal entrance (acute or chronic)
* Status post-tympanoplasty type I-III <3 months
* Acute febrile state
* Optic neuritis
* Unstabilized hyperthyroidism

Contra-indication to MRI :

* Non-MRI-compatible pacemaker, cochlear implant, drug-infusion pump or neurostimulator.
* Metallic foreign body in critical area (eye, brain, etc.)
* Ferromagnetic vascular surgical clips of older generation, e.g., for intracranial aneurysm repair.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of fat graft volume retained | From enrollment until six months after the second lipofilling procedure.
  Fat graft volume retention in % is assessed by comparing preoperative and six-month postoperative MRI measurements.

SECONDARY OUTCOMES:
Absolute retention of fat graft volume | Participants will be followed from enrollment to six months after the second lipofilling procedure.
  Six months after each lipofilling procedure, an MRI is performed to evaluate the absolute retention of fat graft volume (in mL) by comparing preoperative and postoperative MRI scans.
Clinical and radiological complications of lipofilling | Outcomes will be assessed from the time of the first lipofilling procedure through six months following the second procedure.
  During follow-up, after each intervention, patients will be assessed for postoperative complications, including infections, hematoma, implant explantation (if applicable), and reoperation. Radiological complications will also be recorded during each MRI, such as the presence of liponecrosis or oil cysts.
Number of Participants with hyperbaric oxygen therapy Related Adverse Events. | Adverse events will be monitored from the initiation of hyperbaric oxygen therapy until six months after the end of the therapy
  All adverse events related to hyperbaric oxygen therapy will be recorded to assess its safety in the context of the study.
  Premature cessation of hyperbaric oxygen therapy, along with the reasons for discontinuation, will be recorded to assess its tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Kalbermatten, MD, PhD, Study Chair — Geneva University Hospitals, Plastic surgery division

IPD SHARING:
Plan to Share IPD: No
In order to protect patient's privacy and data.

REFERENCES:
- [Background] Strong AL, Cederna PS, Rubin JP, Coleman SR, Levi B. The Current State of Fat Grafting: A Review of Harvesting, Processing, and Injection Techniques. Plast Reconstr Surg. 2015 Oct;136(4):897-912. doi: 10.1097/PRS.0000000000001590. PMID 26086386
- [Background] Andre-Levigne D, Modarressi A, Pignel R, Bochaton-Piallat ML, Pittet-Cuenod B. Hyperbaric oxygen therapy promotes wound repair in ischemic and hyperglycemic conditions, increasing tissue perfusion and collagen deposition. Wound Repair Regen. 2016 Nov;24(6):954-965. doi: 10.1111/wrr.12480. Epub 2016 Oct 18. PMID 27684570
- [Background] Moen I, Stuhr LE. Hyperbaric oxygen therapy and cancer--a review. Target Oncol. 2012 Dec;7(4):233-42. doi: 10.1007/s11523-012-0233-x. Epub 2012 Oct 2. PMID 23054400
- [Background] Meier EL, Mink van der Molen DR, Lansdorp CA, Batenburg MCT, van der Leij F, Verkooijen HM, Boonstra O, Hummelink S, Ulrich DJO. Hyperbaric oxygen therapy for local late radiation toxicity in breast cancer patients: A systematic review. Breast. 2023 Feb;67:46-54. doi: 10.1016/j.breast.2022.12.009. Epub 2022 Dec 22. PMID 36587606
- [Background] De Wolde SD, Hulskes RH, Weenink RP, Hollmann MW, Van Hulst RA. The Effects of Hyperbaric Oxygenation on Oxidative Stress, Inflammation and Angiogenesis. Biomolecules. 2021 Aug 14;11(8):1210. doi: 10.3390/biom11081210. PMID 34439876
- [Background] Liang J, Sun X, Yi L, Lv J. Effect of Hyperbaric Oxygen Therapy on the Survival Rate of Autologous Fat Transplantation. Aesthetic Plast Surg. 2023 Feb;47(1):423-429. doi: 10.1007/s00266-022-03096-y. Epub 2022 Sep 27. PMID 36168069
- [Background] El-Sabawi B, Carey JN, Hagopian TM, Sbitany H, Patel KM. Radiation and breast reconstruction: Algorithmic approach and evidence-based outcomes. J Surg Oncol. 2016 Jun;113(8):906-12. doi: 10.1002/jso.24143. Epub 2016 Jan 11. PMID 26750435
- [Background] Pu LL. Mechanisms of Fat Graft Survival. Ann Plast Surg. 2016 Feb;77 Suppl 1:S84-6. doi: 10.1097/SAP.0000000000000730. PMID 26808753
- [Background] Herly M, Orholt M, Larsen A, Pipper CB, Bredgaard R, Gramkow CS, Katz AJ, Drzewiecki KT, Vester-Glowinski PV. Efficacy of breast reconstruction with fat grafting: A systematic review and meta-analysis. J Plast Reconstr Aesthet Surg. 2018 Dec;71(12):1740-1750. doi: 10.1016/j.bjps.2018.08.024. Epub 2018 Sep 4. PMID 30245019
- [Background] Shim YH, Zhang RH. Literature Review to Optimize the Autologous Fat Transplantation Procedure and Recent Technologies to Improve Graft Viability and Overall Outcome: A Systematic and Retrospective Analytic Approach. Aesthetic Plast Surg. 2017 Aug;41(4):815-831. doi: 10.1007/s00266-017-0793-3. Epub 2017 Feb 7. PMID 28175966
- [Background] Gentilucci M, Mazzocchi M, Alfano C. Effects of Prophylactic Lipofilling After Radiotherapy Compared to Non-Fat Injected Breasts: A Randomized, Objective Study. Aesthet Surg J. 2020 Sep 14;40(10):NP597-NP607. doi: 10.1093/asj/sjaa182. PMID 32598447
- [Background] Batenburg MCT, Maarse W, van der Leij F, Baas IO, Boonstra O, Lansdorp N, Doeksen A, van den Bongard DHJG, Verkooijen HM. The impact of hyperbaric oxygen therapy on late radiation toxicity and quality of life in breast cancer patients. Breast Cancer Res Treat. 2021 Sep;189(2):425-433. doi: 10.1007/s10549-021-06332-2. Epub 2021 Jul 19. PMID 34279734
- [Background] Mink van der Molen DR, Batenburg MCT, Maarse W, van den Bongard DHJG, Doeksen A, de Lange MY, van der Pol CC, Evers DJ, Lansdorp CA, van der Laan J, van de Ven PM, van der Leij F, Verkooijen HM. Hyperbaric Oxygen Therapy and Late Local Toxic Effects in Patients With Irradiated Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2024 Apr 1;10(4):464-474. doi: 10.1001/jamaoncol.2023.6776. PMID 38329746
- [Background] Pandey K, Teguh DN, van Hulst RA. Effect of hyperbaric oxygen treatment on skin elasticity in irradiated patients. Diving Hyperb Med. 2022 Sep 30;52(3):208-212. doi: 10.28920/dhm52.3.208-212. PMID 36100932
- See also: Informative brochure from the Hyperbaric Medicine Division of the Geneva University Hospitals (in French) — https://www.hug.ch/sites/interhug/files/documents/medecine_hyperbare.pdf
- See also: Official website of the Hyperbaric Medicine Division of the Geneva University Hospitals with an explanatory video — https://www.hug.ch/programme-medecine-hyperbare/deroulement-traitement